CLINICAL TRIAL: NCT04450251
Title: Testing a Wearable Monitor for Fetal Heart Rate Estimation, Fetal
Brief Title: Testing a Wearable Monitor for Fetal Heart Rate Estimation, Fetal Movement and Uterine Activity Detection
Status: Completed | Type: Observational
Sponsor: Owlet Baby Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OWLET-01
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy
Keywords: Pregnancy Tracker; Owlet Band; Owlet; Wearable Tech
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women, at least 24 weeks gestation
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Collect observational fetal electrocardiogram (ECG) readings with a novel wearable device.

SUMMARY:
Owlet Baby Care, Inc. has developed a wearable fabric band pregnancy monitor, to be worn around the maternal abdomen incorporating electrocardiogram sensors. The purpose of this proposed test is to collect overnight "at-home" fetal ECG recordings on women during the second half of pregnancy using the pregnancy monitor.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman, 18 years of age and up.
* Singleton or twin pregnancy.

Exclusion Criteria:

* Self-reported substance abuse problems.
* Anyone unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 500 pregnant women 24 weeks gestation and up in the second or third trimester of pregnancy will be screened into the study.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to collect observational fetal ECG readings with a novel wearable device | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ward, MD, Principal Investigator — Owlet Baby Care, Inc.
Locations (1):
- Owlet Baby Care, Inc., Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No